CLINICAL TRIAL: NCT05697549
Title: Effects of Cognitive Behavior Language Therapy for Patients With Post Stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: aleena1irum
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cognitive behavior language therapy (Experimental): Cognitive behavior language therapy is an extensive form of CBT. And it is focused on the treatment of speech-language related problems. CBLT helped the individuals to change their unhelpful thoughts and beliefs that cause difficulty for them to communicate properly and effectively. The main aim of CBLT is to use their remaining language abilities, to restore their language abilities and to learn the other ways of communication i.e. pointing, gesturing and AAC.
  Interventions: Behavioral: cognitive behavior language therapy

INTERVENTIONS:
Behavioral: cognitive behavior language therapy — Cognitive behavior language therapy is an extensive form of Cognitive behavior therapy. and it is used in the management of speech-language related problems. It helps the individuals to change their unhelpful thoughts and beliefs that cause difficulty for them to communicate properly and effectively. and it also helps the individuals to use their remaining language abilities, to restore their language abilities and to learn the other ways of communication i.e. pointing, gesturing and Augmentative alternative communication.

SUMMARY:
This study is clinical trial based and the target population in this study is patients with post-stroke aphasia. Cognitive linguistic quick test (CLQT) and Speech Language unhelpful thoughts and belief scale (SLUTBS) will apply as an assessment. Inclusive criteria include diagnosed male and female post-stroke severe aphasia patients above 30 years of age. These participants must have high instance of unhelpful speech language thoughts and belief. Participants in inclusive criteria must not be participated in any other psychotherapy/ speech language intervention program. Participants must sign an informed consent form. Participants having a caregiver who is willing to be present during the period of intervention. Exclusive criteria include individuals below 30 years of age and patients with aphasia caused by non-stroke etiology.

The aim of the study is to check the effects of cognitive behavior language therapy on patients with post-stroke aphasia. So, it will help speech language pathologists to adopt the principles of CBLT intervention to treat aphasia that occurs as a result of aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female.
* Over 30 years of age.
* All types of diagnosed aphasia.
* Severe aphasia following stroke.
* High instance of unhelpful speech language thoughts and belief.
* Participants who are not participating in any other psychotherapy / speech language intervention program will be included.
* Participants who are willing to sign an informed consent form.
* Participants having a caregiver who is willing to be present during the period of intervention.

Exclusion Criteria:

* Below 30 years of age.
* Patients with aphasia caused by a non-stroke etiology.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — both male and female will be included.
Enrollment: 30 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Cognitive linguistic quick test | 4 week
  scoring 3.5 to 4 indicates attention, memory, executive functions, language, visuospatial skills are within the normal limit. whereas scoring 1 to 1.4 indicates that individual has severely affected in these areas.
Speech language and helpful thoughts and belief scale | 4 week
  the scoring of this scale according to 4. Likert scale. In which ''4'' strongly agree indicates high communication gap while sharing thoughts with others and ''1'' strongly disagree indicates individuals haven't facing any difficulties while sharing thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Aleena Irum, MSLP, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zaid, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No